CLINICAL TRIAL: NCT03696602
Title: More Relaxation by Deep Breath on Methacholine- Than on Exercise-Induced Bronchoconstriction During the Routine Testing of Asthmatic Children
Brief Title: More Relaxation by Deep Breath on Methacholine
Acronym: SouProvocBro
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: enf4327
Record Dates: First submitted 2018-09-21; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Childhood Asthma
Keywords: airway smooth muscle, asthma, bronchial test, lung function
MeSH Terms: conditions — Asthma | interventions — Bronchial Provocation Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test with methacholine
  Interventions: Diagnostic Test: bronchial provocation test
- test with exercise
  Interventions: Diagnostic Test: bronchial provocation test

INTERVENTIONS:
Diagnostic Test: bronchial provocation test

SUMMARY:
Deep inhalation (DI) dilates normal airway precontracted with methacholine. The fact that this effect is diminished or absent in asthma could be explained by the presence of bronchial inflammation. The hypothesis tested was that DI induces more relaxation in methacholine induced bronchoconstriction-solely determined by the smooth muscle contraction-than in exercise induced bronchoconstriction, which is contributed to by both smooth muscle contraction and airway wall inflammation.

DETAILED DESCRIPTION:
Children were referred to the lung function department by their pediatric pulmonologist. Asthma was defined by a complaint of wheezing, cough, dyspnoea or chest tightness at rest or on exercising and a positive response to methacholine or exercise challenge.

The response to exercise was considered positive when Forced Expiratory Volume in 1 s (FEV1) decreased at least 8% from Baseline.

The response to methacholine was considered positive when FEV1 decreased at least 20% or Rrs increased at least 50% from baseline, at or below a cumulated dose of 1,200 μg.

Bronchodilator medications were discontinued at least 12 hours prior to the testing and provocation allowed when the child had been free of respiratory symptoms for at least 2 weeks and baseline FEV1 was larger than 70% pred. Exercise and methacholine groups were matched for age, height, baseline FEV1 z-score, a moderate level of airway response to challenge and DI amplitude ranging 40-60% of the predicted Forced Vital Capacity (FVC). Written informed consent was obtained from the children and their parents for the procedures. Procedures for spirometry, exhaled fraction of NO (FENO), GrsDI (Respiratory conductance response to a deep inhalation) and challenges have been described previously. Acceptable GrsDI's were analyzed at a 10-20% FEV1 decrease from baseline. Statistics were performed using Mann-Whitney, Chi square tests and multiple regression as required. Data are median and interquartile range.

ELIGIBILITY:
Inclusion Criteria:

* Children referred to the lung function department by their pediatric pulmonologist.
* Asthma defined by a complaint of wheezing, cough and dyspnoea.
* Positive response to methacholine or exercise challenge.
* Bronchodilator medications discontinued at least 12 h prior to the testing
* Provocation allowed when the child had been free of respiratory symptoms for at least 2 weeks and baseline FEV1 larger than 70% pred.

Exclusion Criteria:

- Other respiratory diseases than asthma

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Seventy-three asthmatic children (48 boys) were selected, 37 underwent exercise challenge and 36 methacholine.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Grs change between before deep breath and after deep breath in exercise and metacholine groups | through study completion, an average of 1 hour
  GrsDI represents Grs measured after deep breath reported to Grs before deep breath (bronchial provocation test)